CLINICAL TRIAL: NCT03774888
Title: A Randomized Controlled Trial to Compare the Histomorphometric and Clinical Outcomes of Soft Tissue Augmentation at the Time of Lateral Ridge Augmentation Procedures
Brief Title: To Compare Different Soft Tissue Grafts at the Time of Lateral Ridge Augmentation Procedure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hussein Basma, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002688
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-11

CONDITIONS: Bone Graft; Complications, Infection or Inflammation; Ridge Deficency; Dental Implant
Keywords: Keratinized Tissue; Keratinized mucosa; attached mucosa; dental implants; ridge augmentation; guided bone regeneration; connective tissue graft; acellular demral matrix
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- connective tissue graft (Experimental): Connective tissue grafting (CTG) will be placed at the time of lateral ridge augmentation.Following the placement of the bone graft and the membrane, a CTG will be harvested and sutured to the membrane and then the flaps passively sutured on top on the bone and soft tissue graft
  Interventions: Procedure: Connective tissue graft at time of bone graft
- Acellular Dermal Matrix (Experimental): Acellular Dermal matrix (ADM) will be placed at the time of lateral ridge augmentation.Following the placement of the bone graft and the membrane, an ADM will be sutured to the membrane and then the flaps passively sutured on top on the bone and soft tissue graft
  Interventions: Procedure: Acellular Demal Matrix at time of bone graft
- No soft tissue graft (Control) (Active Comparator): Control group where no soft tissue graft is added to the lateral ridge augmentation.Following the placement of the bone graft and the membrane, the flaps passively sutured on top on the bone. No soft tissue graft will be added.
  Interventions: Procedure: No soft tissue grafting at time of bone graft

INTERVENTIONS:
Procedure: Connective tissue graft at time of bone graft — following the placement of the bone graft and the membrane, a CTG will be harvested and sutured to the membrane and then the flaps passively sutured on top on the bone and soft tissue graft
  Arms: connective tissue graft
Procedure: Acellular Demal Matrix at time of bone graft — following the placement of the bone graft and the membrane, an ADM will be sutured to the membrane and then the flaps passively sutured on top on the bone and soft tissue graft
  Arms: Acellular Dermal Matrix
Procedure: No soft tissue grafting at time of bone graft — Following the placement of the bone graft and the membrane, the flaps passively sutured on top on the bone. No soft tissue graft will be added.
  Arms: No soft tissue graft (Control)

SUMMARY:
This study will compare two commonly used soft tissue grafting techniques (connective tissue graft, CTG vs Acellular Dermal Matrix, ADM) to augment the soft tissue at the time of lateral ridge augmentation procedure.

Following ridge augmentation procedure, most of the times there is a need for soft tissue augmentation to change the quality of the tissue around future implant's site. To our knowledge, the influence of soft tissue augmentation at the time of ridge augmentation procedure has not been tested defects.

DETAILED DESCRIPTION:
Research data and daily clinical observations reveal that implants with lack of surrounding keratinized mucosa KM (gingiva-like tissue that normally surrounds natural teeth) are more prone to persistent gingival inflammation, faster disease progression and compromised plaque control. Ridge augmentation procedure can alter the quality of tissue in the sites where it will receive dental implants. Soft tissue grating aims at changing the nature of peri-implant soft tissue by creating or increasing the zone of keratinized mucosa (KM) surrounding implants. CTG or ADM will be grafted at the same time of lateral ridge augmentation procedure.

Specific aims for this project include the evaluation of:

1. To evaluate the quality of soft tissue regenerated with the use of the two available soft tissue grafts via histological analysis.
2. To evaluate whether CTG or ADM influences the outcomes of Guided Bone Regeneration (GBR) procedures.
3. To quantify the soft tissue augmentation achieved by the two available soft tissue grafts by direct clinical measurements after the healing

ELIGIBILITY:
Inclusion Criteria:

1. Be a registered University of Alabama at Birmingham (UAB) dental school patient
2. English Speaking
3. Healthy enough to undergo the proposed therapy
4. Demonstrated willingness to comply with study directions and time-line
5. Insufficient alveolar ridge width for endosseous implant placement defined as 5mm or less as determined by bone sounding and cone beam computed tomography (CBCT) scan.
6. Able to read and understand the informed consent form
7. Need for implants to replace missing tooth or teeth in at least one quadrant of the mouth.

Exclusion Criteria:

1. No English Speaking
2. Smokers/ tobacco users (>10 cigarettes a day)
3. Less than 18 years old
4. Know hypersensitivity to titanium
5. Patients with significant medical conditions or habbits expected to interfere with bony healing.
6. Patient is a poor compliance risk (i.e., poor oral hygiene, history of alcohol or drug abuse)
7. Bone dehiscence of >4mm following tooth extraction or Vertical loss of bone at edentulous ridge

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Basma, DDS, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Unversity of Alabama at Birmingham, School of Dentistry, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in the School of Dentistry Periodontology Clinic in need of grafting treatment will be told about the study and if interested in participation will be scheduled for a screening visit for study entry by periodontal residents and faculty members.
  Randomization was performed by site in the mouth (dental implant site) to receive either CTG intervention, ADM or control. Total CTG sites=13, total ADM sites=16 and control sites=12.
Units Other Than Participants: dental implant site
Period: Overall Study
Arm/Group | Connective Tissue Graft | Acellular Dermal Matrix | No Soft Tissue Graft (Control)
Started | 8; 13 dental implant site | 8; 16 dental implant site | 8; 12 dental implant site
Completed | 8; 13 dental implant site | 8; 16 dental implant site | 8; 12 dental implant site
Not Completed | 0; 0 dental implant site | 0; 0 dental implant site | 0; 0 dental implant site

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Connective Tissue Graft | Acellular Dermal Matrix | No Soft Tissue Graft (Control) | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 4 | 13
  >=65 years | 2 | 5 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 7 | 15
  Male | 5 | 3 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 6 | 7 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 7 | 7 | 8 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Measure Changes Clinically in Crestal Soft Tissue Thickness (in mm)
Description: The changes in clinical vertical crestal soft tissue thickness by using an endodontic file and periodontal probe.
Time Frame: From baseline to 6 months
Population: Randomization was performed by site in the mouth (dental implant site) to receive either CTG intervention, ADM or control. Total CTG sites=13, total ADM sites=16 and control sites=12.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: dental implant site
Arm/Group | Connective Tissue Graft | Acellular Dermal Matrix | No Soft Tissue Graft (Control)
Number analyzed (Participants) | 8 | 8 | 8
Number analyzed (dental implant site) | 13 | 16 | 12
mm | 1.96 (1.05) | 1.59 (1.06) | 0.33 (1)

2. Primary Outcome: Measure Changes Digitally in Crestal Soft Tissue Thickness (in mm)
Description: The changes in soft tissue thickness digitally with superimposition of the intraoral scan and cone-bone computed tomography scan.
Time Frame: From baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: dental implant site
Arm/Group | Connective Tissue Graft | Acellular Dermal Matrix | No Soft Tissue Graft (Control)
Number analyzed (Participants) | 8 | 8 | 8
Number analyzed (dental implant site) | 13 | 16 | 12
mm | 1.65 (0.95) | 0.74 (0.93) | -0.09 (0.61)

3. Primary Outcome: Measure Changes Clinically in Soft Tissue Thickness at 4mm Apical From Gingival Margin
Description: The changes in clinical soft tissue thickness at 4mm apical form the gingival margin by using an endodontic file and periodontal probe.
Time Frame: From baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: dental implant site
Arm/Group | Connective Tissue Graft | Acellular Dermal Matrix | No Soft Tissue Graft (Control)
Number analyzed (Participants) | 8 | 8 | 8
Number analyzed (dental implant site) | 13 | 16 | 12
mm | 2.38 (1.32) | 1.37 (1.2) | 0.15 (1.65)

4. Primary Outcome: Measure Changes Digitally in Soft Tissue Thickness at 4mm Apical Form Gingival Margin
Description: as for outcome 2
Time Frame: From baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: dental implant site
Arm/Group | Connective Tissue Graft | Acellular Dermal Matrix | No Soft Tissue Graft (Control)
Number analyzed (Participants) | 8 | 8 | 8
Number analyzed (dental implant site) | 13 | 16 | 12
mm | 1.75 (0.87) | 1.23 (0.7) | 0.71 (0.57)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | Connective Tissue Graft | Acellular Dermal Matrix | No Soft Tissue Graft (Control)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Randomization was performed by site (dental implant) due to challenges recruiting sufficient participants for all arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03774888/Prot_SAP_000.pdf